CLINICAL TRIAL: NCT02927223
Title: Pretreatment With Atropine to Reduce Exercise-triggered Ventricular Ectopy in Patients With Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Brief Title: Atropine in Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Prince Joseph Kannankeril, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VUMC-161398
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia
MeSH Terms: conditions — Polymorphic Catecholaminergic Ventricular Tachycardia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treadmill then Treadmill with Atropine (Experimental): Patients will undergo treadmill exercise at baseline, then Patients will undergo treadmill exercise after IV atropine
  Interventions: Drug: Atropine; Procedure: Exercise treadmill test

INTERVENTIONS:
Drug: Atropine
Procedure: Exercise treadmill test

SUMMARY:
To test the hypothesis that increasing the sinus node rate with atropine treatment prior to exercise will reduce exercise-triggered ventricular ectopy compared to baseline in patients with CPVT.

DETAILED DESCRIPTION:
This is a prospective cross-over trial that will enroll eligible patients with CPVT and perform a baseline treadmill exercise tolerance test (ETT) followed by a repeat treadmill ETT with I.V. atropine administered immediately prior to exercise. Atropine is a parasympathetic blocker and results in sinus tachycardia, which is expected to reduce the diastolic interval thereby reducing delayed after depolarizations and ventricular ectopy compared to baseline. Both ETTs will be performed on the same day with two hours of rest scheduled between ETTs. The primary analysis will be a paired comparison of the number of ventricular ectopic beats recorded during exercise (and recovery) at baseline and following pre-treatment with atropine. Secondary endpoints will include the presence of ventricular ectopy (yes/no), complex ventricular ectopy (couplets or greater, yes/no), and the number of runs of complex ventricular ectopy.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 6 years
* Able to provide written informed consent
* Clinical diagnosis of CPVT
* Able to exercise on a treadmill
* Successful completion of a minimum of 2 exercise stress tests without adverse events

Exclusion Criteria:

* Contraindication to treadmill stress testing according to Vanderbilt University Medical Center's clinical protocols (unstable angina, decompensated congestive heart failure, severe hypertension (≥ 170/90 mmHg), acute myocardial infarction (<4 days), moderate to severe aortic stenosis, acute pulmonary embolism, severe pulmonary hypertension, outflow tract obstruction, hypertrophic cardiomyopathy, left main coronary stenosis, left bundle branch block)
* Females who are pregnant
* In the judgement of the investigator, any clinically significant ongoing medical or surgical condition that might jeopardize the subject's safety or interfere with the conduct of the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prince J Kannankeril, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kannankeril PJ, Shoemaker MB, Gayle KA, Fountain D, Roden DM, Knollmann BC. Atropine-induced sinus tachycardia protects against exercise-induced ventricular arrhythmias in patients with catecholaminergic polymorphic ventricular tachycardia. Europace. 2020 Apr 1;22(4):643-648. doi: 10.1093/europace/euaa029. PMID 32091590

RESULTS

PARTICIPANT FLOW:
Groups:
- Treadmill Then Treadmill With Atropine: Patients will undergo treadmill exercise at baseline, then Patients will undergo treadmill exercise after IV atropine
  Atropine
  Exercise treadmill test
Period: Overall Study
Arm/Group | Treadmill Then Treadmill With Atropine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treadmill Then Treadmill With Atropine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 38 [22 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventricular Ectopic Beats Recorded During Exercise (and Recovery)
Time Frame: 20 minutes during exercise
Measure: Median (Full Range); unit: number of ventricular beats
Groups:
- Treadmill: Patients will undergo treadmill exercise at baseline,
  Exercise treadmill test
- Treadmill With Atropine: Patients will undergo treadmill exercise after IV atropine
  Atropine
  Exercise treadmill test
Arm/Group | Treadmill | Treadmill With Atropine
Number analyzed (Participants) | 6 | 6
number of ventricular beats | 46 [6 to 192] | 0 [0 to 29]

ADVERSE EVENTS:
Time Frame: 7 hours
Arm/Group | Treadmill | Treadmill With Atropine
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02927223/Prot_SAP_001.pdf